CLINICAL TRIAL: NCT03157414
Title: Efficacy and Safety of Empagliflozin in Renal Transplant Recipients With Post-transplantation Diabetes Mellitus
Brief Title: Empagliflozin in Renal Transplant Recipients
Acronym: EMPA-RenalTx
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Trond Jenssen, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016/911; 2016-001705-17 (EudraCT Number); 2016069 (Other Grant/Funding Number: South-Eastern Norway Regional Health Authority)
Record Dates: First submitted 2017-03-15; First posted 2017-05-17 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus; Renal Insufficiency; Safety Issues
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Active Comparator): 10 mg once daily for 24 weeks
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): 1 capsule once daily for 24 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin tablets enclosed with red capsules (Capsugel AAEL) by Kragerø Tablettproduksjon AS for blinding purpose
  Other Names: Jardiance
  Arms: Empagliflozin
Other: Placebo — Placebo tablets made by Kragerø Tablettproduksjon AS and enclosed with red capsules (Capsugel AAEL) for blinding purpose
  Arms: Placebo

SUMMARY:
This is a single-center, prospective, controlled, double-blind, randomized study. A total of 50 renal transplant recipients diagnosed with post-transplantation diabetes mellitus (PTDM) will be included more than 1 year after transplantation and randomized 1:1 to empagliflozin (Jardiance®) 10 mg or placebo once daily for 24 weeks. Patients with estimated glomerular filtration rate below 30 mL/min will be excluded. Oral glucose tolerance test, 72h continuous glucose monitoring (iPro™2), measurement of arterial stiffness, body composition (including visceral fat), 24h blood pressure and 24h urinary glucose excretion will be performed at baseline and after 24 weeks in addition to standard safety measurements. Two safety visits will be performed at week 8 and 16. All concomitant medication, diet and exercise will be kept stable during the study period. The objective of the present study is to answer whether empagliflozin safely and effectively improves glucose metabolism together with weight loss in renal transplant recipients with PTDM.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipient transplanted more than 1 year ago
* Stable renal function (<20% deviation in serum creatinine within last 2 months)
* Stable immunosuppressive therapy ≥3 months before inclusion
* Diagnosed with PTDM:

(fasting plasma glucose ≥7.0 mmol/l and/or 2-hour plasma glucose ≥11.1 mmol/l following an oral glucose tolerance test)

-Signed informed consent and expected cooperation of the patients

Exclusion Criteria:

* Estimated GFR <30 ml/min/1.73 m2
* Pregnant or nursing mothers
* Hypersensitivity to the active substance (IMP) or to any of the excipients
* Any reason why, in the opinion of the investigator, the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Weighted mean glucose | 24 weeks
  The primary endpoint will be change from baseline in weighted mean glucose at week 24 compared to placebo. Each patient will perform continuous plasma glucose monitoring (CGM, iProTM2) for 72 hours at baseline and after 24 weeks.

SECONDARY OUTCOMES:
Fasting plasma glucose | 24 weeks
  Change from baseline in fasting plasma glucose
2 hour glucose concentration | 24 weeks
  Change from baseline in 2 hour glucose concentration after an oral glucose tolerance test
Glycated hemoglobin (HbA1c) | 24 weeks
  Change from baseline in HbA1c
Body weight | 24 weeks
  Change from baseline in body weight
Waist-hip-ratio | 24 weeks
  Change from baseline in waist-hip-ratio
Bone mineral density | 24 weeks
  Measurement of bone mineral density, using low dosage radiation (dual-energy X-ray absorptiometry (DEXA) scan) to assess the amount (grams) of mineral that are packed into a segment of bone
Body composition | 24 weeks
  Body composition (visceral fat, metabolic measurement) will be determined using the software CoreScan (encore version 14.10, GE Healthcare) on the DEXA scans. This will allow us to analyze changes in body fat compartments to explain overall weight reduction
Blood pressure | 24 weeks
  Change from baseline in blood pressure, including orthostatic blood pressure
Arterial stiffness | 24 weeks
  Pulse wave velocity, using a SphygmoCor device, measuring arterial stiffness will be performed in addition to pulse wave analysis evaluating the shape and amplitude of the aortic pulse wave
Renal function | 24 weeks
  Renal function, defined as glomerular filtration rate (GFR), will be evaluated by creatinine and cystatin C-based estimated GFR using the chronic kidney disease epidemiology collaboration (CKD-EPI) formula. Fasting plasma creatinine and Cystatin C will be drawn at the same time and analyses will be performed at the Hospital central laboratory

OTHER OUTCOMES:
Incidence of abnormal trough levels of immunosuppressive drugs | 24 weeks
  Trough levels of immunosuppressive drugs (tacrolimus); number of participants with abnormal laboratory values
Adverse event | 24 weeks
  Recording of adverse events that are related to treatment
Urinary glucose excretion | 24 weeks
  24 hour urine sampling at baseline and after 24 weeks to analyse change in urinary glucose excretion

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lo C, Toyama T, Oshima M, Jun M, Chin KL, Hawley CM, Zoungas S. Glucose-lowering agents for treating pre-existing and new-onset diabetes in kidney transplant recipients. Cochrane Database Syst Rev. 2020 Jul 30;8(8):CD009966. doi: 10.1002/14651858.CD009966.pub3. PMID 32803882
- [Derived] Halden TAS, Kvitne KE, Midtvedt K, Rajakumar L, Robertsen I, Brox J, Bollerslev J, Hartmann A, Asberg A, Jenssen T. Efficacy and Safety of Empagliflozin in Renal Transplant Recipients With Posttransplant Diabetes Mellitus. Diabetes Care. 2019 Jun;42(6):1067-1074. doi: 10.2337/dc19-0093. Epub 2019 Mar 12. PMID 30862658